# Analyzing the Patterns of Patient Engagement and Trends in Participation Observed in Medullary Thyroid Cancer Clinical Trials

This is an Informed Consent Form For Medullary Thyroid Cancer Patients in <a href="Power Clinical Trial's">Power Clinical Trial's</a> Observational Study

Date: October 6, 2023

Comprehending the Significance of This Consent Form

If you find yourself completing this document, it indicates your potential eligibility for participation in a unique observational clinical study dedicated to medullary thyroid cancer patients. This comprehensive guide outlines the study's core goals, intricate implementation plan, and various implications, encompassing both positive and potentially adverse outcomes. Prior to making a decision, it is imperative to thoroughly investigate the specifics of your potential participation, and seeking counsel from a trusted source can offer valuable perspectives. Should any part of this text appear confusing or if you have questions, know that the researcher is available to provide clarification.

Recognizing the Importance of Medullary Thyroid Cancer Clinical Trials

Medullary thyroid cancer (MTC) is a rare type of thyroid cancer that originates in the parafollicular C cells of the thyroid gland. These C cells are responsible for producing a hormone called calcitonin, which helps regulate calcium levels in the body. Unlike the more common types of thyroid cancer (such as papillary and follicular thyroid cancer), which arise from thyroid hormone-producing cells, MTC arises from these distinct C cells.

Clinical studies, with a distinct emphasis on medullary thyroid cancer, play a pivotal role in evaluating the safety and effectiveness of novel treatments for this condition. These trials serve as essential tools to determine whether new medications surpass conventional therapies, providing substantial evidence to endorse their broader adoption.

What sets this particular study apart is its central focus on the firsthand experiences of individuals dealing with medullary thyroid cancer, actively participating in a clinical trial incorporating medicinal interventions. The primary objective is to meticulously examine trial completion rates and voluntary withdrawals within this specific patient group.

# **Exploring the Essence of Observational Clinical Trials**

Participating in this medical trial entails being immersed in an observational study, a distinct element of clinical research that is precisely designed to gather insights through unobtrusive monitoring of patients while maintaining their treatment regimens.

Researchers will just monitor your trip, meticulously assessing the results of your condition and make no changes. This particular trial design is critical in improving our understanding of the underlying evolution of a certain medical disease and its consequences for those affected by it. By actively participating in this observational study, you play a critical role in pushing medical knowledge forward and advancing care for individuals suffering from the same problem.

This Study As Distinguished From Other Medullary Thyroid Cancer Clinical Trials

It is critical to recognize the unique elements of this research investigation. It is entirely observational, which means that your participation will not entail any particular therapies or interventions. To make an educated choice about prospective participation in a clinical trial, it is critical to understand the range of medullary thyroid cancer clinical research, including interventional studies in which participants receive a variety of treatment regimens.

Making an informed decision regarding your future involvement in a clinical trial necessitates an active approach that includes research and trial comparison. Clinicaltrials.gov and other comparable sites include a plethora of information about

<u>medullary thyroid cancer research</u>. Power's dedicated online platform also provides a complete list of ongoing <u>medullary thyroid cancer clinical trials</u> that are actively seeking volunteers. Armed with meticulous study and a thorough comprehension of several clinical trial categories, you may define your participation decision firmly.

# Ensuring the Security of Your Answers

During the course of this research project, it is critical to ensure the total confidentiality of your data. To protect your anonymity, please do not include any personal or identifiable information in your questionnaire replies. The committed research team is steadfast in their quest to strengthen your privacy protection. Nonetheless, it is critical to recognize that some legal conditions may emerge that necessitate the sharing of personal data.

# Actively Contributing to Clinical Trial Surveys: Your Voice Matters

We cordially invite you to actively share your experiences within the context of this observational clinical study. This initiative entails completing surveys every two weeks, which will take around 20-30 minutes of your valuable time. Furthermore, we are well prepared to conduct quarterly check-in calls, a practice that will continue during your participation in the trial.

It is critical to underline that your participation in the trial's survey phase is totally voluntary. You have the option of responding to individual questions or completing the full questionnaire. Furthermore, you have the option to withdraw from the trial at any time if you so want. Recognizing that enrolling in a clinical trial is a very personal decision, we are committed to providing the appropriate assistance. We value your privacy and comfort, and we are devoted to respecting and aiding you in making decisions during the trial.

# **Expectations of Potential Benefits**

While participants in this observational clinical research may not see immediate advantages, their participation has the potential to have a significant impact on others. The information gathered from participants will be used to enhance future tactics for recruiting people with medullary thyroid cancer, potentially broadening the scope of

medical research. Those who embark on this treatment journey have the potential to spark substantial changes in medical research, perhaps paving the way for future medullary thyroid cancer sufferers.

# Recognizing Potential Health Consequences

While clinical trials have resulted in tremendous progress, it is critical to recognize the possible health risks that participants may suffer, especially in studies assessing new drugs.

However, our technique in observational clinical research takes a unique approach, limiting these disadvantages by not administering experimental medicines to subjects. Instead, our major focus is on extensive monitoring and outcome evaluation, assuring the avoidance of any unnecessary health hazards.

# Empowering Diversity in Clinical Investigations

Numerous internet routes anxiously await your active participation if you are driven by an insatiable passion to investigate the multidimensional element of diversity in clinical trials.

Whether your objective is to get an understanding of the nuances of the issues and possibilities related to clinical trial diversity or to broaden your own viewpoints, the following materials might be quite useful:

Clark, Luther T., Laurence Watkins, Ileana L. Piña, Mary Elmer, Ola Akinboboye, Millicent Gorham, Brenda Jamerson et al. "Increasing diversity in clinical trials: overcoming critical barriers." *Current problems in cardiology* 44, no. 5 (2019): 148-172.

Knepper, Todd C., and Howard L. McLeod. "When will clinical trials finally reflect diversity?." (2018): 157-159.

### Validation of Informed Consent

I certify that I have spent sufficient time understanding and internalizing the information included in the informed consent form. This understanding has come from either

independent research or the direction of a trusted someone who has explained its contents to me. All of my issues and inquiries have been thoroughly answered to my great satisfaction.

I am fully aware that my participation in this study is entirely voluntary, and I maintain the only right to withdraw my permission without being required to present reasons or take financial responsibility. I have been assured that I will receive a copy of this informed consent form for my own records.

I thus grant my agreement to participate in this study after careful deliberation and a comprehensive assessment of the information supplied to me, indicating my informed and autonomous decision.

| Participant Name |
|-----------------------|
| · |
| Participant Signature |
| Date |

# Confirmation by Informed Consent Facilitator

I affirm that I had a thorough discussion with the participant, thoroughly clarifying the complexities included within this written document. My goal was to ensure that the participant had a complete grasp of the major study goals, methods used, potential risks and rewards, and other important aspects of the medullary thyroid cancer clinical trial.

The participant had enough chances to ask questions, voice concerns, and seek clarification. It is critical to emphasize that participants' participation in this study is fully voluntary, and they have the unrestricted right to leave at any time, for any reason, without incurring any financial responsibilities.

| Following the participant's assent, they we this written document, which served as a | ere given a meticulously preserved replica of repository for their personal information. |
|---|---|
| Printed Name of Assisting Researcher | |
| Signature of Assisting Researcher | |
| Date | |